CLINICAL TRIAL: NCT06362590
Title: Expanded Access Use of Ladiratuzumab Vedotin in Advanced Solid Tumors
Status: Available | Type: Expanded Access
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LV-SPIND-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ladiratuzumab vedotin

SUMMARY:
The purpose of this study is to provide the option of Ladiratuzumab Vedotin treatment to eligible patients in studies SGNLVA-005.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult